CLINICAL TRIAL: NCT06983405
Title: Effectiveness of a Physical Therapy Program Based on Therapeutic Physical Exercise and Health Education to Improve Quality of Life and Health Status in Major Depressive Disorder: A Mixed-Method Pilot Study Protocol
Brief Title: Physical Therapy for Depression Quality of Life (Pilot Study Protocol)
Acronym: PTEduQoL-MDD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad San Jorge (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 38/3/24-25
Record Dates: First submitted 2025-04-24; First posted 2025-05-21 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Major Depressive Disorder (MDD)
Keywords: Major Depressive Disorder; Physical Therapy; Therapeutic Exercise; Health Education; Pilot Study; Quality of Life; Mental Health
MeSH Terms: conditions — Depressive Disorder, Major; Health Education; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: This pilot study employs a concurrent nested mixed-methods design. One group of participants will consist of adult patients admitted to the short-stay psychiatric unit diagnosed with Major Depressive Disorder. This patient group will participate in both the quantitative phase, involving pre- and post-intervention assessments of quality of life, depressive symptoms, and self-efficacy, and the qualitative phase, participating in focus groups to explore their experiences and perceptions. A separate group of participants will comprise healthcare professionals (including medical, nursing, and other allied health staff) working in the same psychiatric unit. This professional group will exclusively participate in the qualitative phase through focus groups to provide their perspectives on the implementation of the physical therapy intervention and its impact on patient management.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Physical Therapy Intervention Group (Experimental): Participants in this arm will receive a physical therapy program consisting of twice-weekly, 45-minute sessions of active joint mobility exercises, strength exercises (body weight/elastic bands), balance exercises, and progressive muscle relaxation, integrated with health education on the relationship between physical activity and mental health, benefits of exercise, strategies for increasing physical activity, self-assessment techniques, and community resources. This intervention will be delivered in addition to their standard medical, psychological, and pharmacological treatment for Major Depressive Disorder.
  Interventions: Other: Physical Therapy Program for MDD

INTERVENTIONS:
Other: Physical Therapy Program for MDD — PT program for hospitalized adults with MDD: twice-weekly, 45-min sessions integrating: 1) Active joint mobility (gentle movements for ROM). 2) Progressive strength (bodyweight/bands, low-mod intensity, major muscles). 3) Balance (stability exercises, adapted difficulty). 4) Progressive muscle relaxation (end of session). Includes health education: exercise & mental health link (biological/psychological mechanisms), benefits of each exercise type (mood, function, QoL), post-discharge activity strategies, self-assessment, community resources in Zaragoza. Delivered by trained PTs, adaptable to individual needs.

SUMMARY:
Major Depressive Disorder (MDD) significantly impacts quality of life and health status. Standard treatments include medical, psychological, and pharmacological approaches, with physical therapy often playing a less central role. This pilot study aims to investigate the potential benefits of incorporating a physical therapy program, based on therapeutic exercise and health education, within the management of MDD in a short-stay psychiatric unit.

This project will implement a physical therapy intervention consisting of twice-weekly sessions of active joint mobility exercises, strength training (body weight/elastic bands), balance exercises, and progressive muscle relaxation, integrated with health education on the benefits of physical activity for mental health and strategies for long-term adherence.

Adult patients (over 18 years) diagnosed with MDD, admitted to the short-stay psychiatry unit of Royo Villanova Hospital in Zaragoza and under regular medical, psychological, and pharmacological treatment, will be recruited for this study. All participants will receive the physical therapy program in addition to their standard care.

The main objective is to analyze the preliminary efficacy of a physical therapy intervention program based on health education and therapeutic exercise in improving quality of life and health status in adults with MDD during their stay in a short-stay psychiatric unit.

A secondary objective is to explore the perceptions of these patients and the healthcare professionals regarding the implementation of this multimodal treatment approach, including barriers and facilitators encountered.

Hypothesis: A physical therapy program integrating therapeutic exercise and health education is feasible and preliminarily effective in improving quality of life and health status in adults with MDD in a short-stay psychiatric unit and is perceived positively by both patients and healthcare professionals regarding its implementation.

DETAILED DESCRIPTION:
This project employs a concurrent nested mixed-methods pilot study with quantitative dominance to evaluate a physical therapy intervention program for adults with Major Depressive Disorder (MDD) within a short-stay psychiatric unit. The quantitative component utilizes a quasi-experimental pre-post design, while the qualitative aspect employs a narrative design through focus groups.

Intervention Protocol:

The physical therapy intervention will be delivered by trained physical therapists in twice-weekly, 45-minute sessions tailored to the participant's length of hospital stay (anticipated 3-6 weeks). Each session will systematically incorporate:

Active Joint Mobility: A series of gentle, controlled movements targeting major joints to maintain or improve their range of motion.

Progressive Strength Training: Low-to-moderate intensity exercises utilizing the participant's own body weight and progressive resistance elastic bands, focusing on key muscle groups.

Balance Enhancement: A structured set of exercises designed to improve stability and reduce the risk of falls, with the difficulty level adapted to each individual's functional capacity.

Relaxation Techniques: Progressive muscle relaxation exercises will be implemented at the conclusion of each session to facilitate physical and mental relaxation.

Integrated Health Education:

Concurrent with the exercise program, participants will receive brief, integrated health education. This component will cover:

The physiological and psychological links between physical activity and mental well-being.

The specific benefits of the exercises within the program concerning mood, physical function, and overall quality of life.

Practical strategies for incorporating and maintaining physical activity as part of their lifestyle post-discharge.

Methods for self-monitoring physical activity levels and mood changes to enhance self-efficacy.

Information regarding available community resources and physical activity programs that participants can access after leaving the hospital.

Qualitative Data Collection Protocol:

Separate focus groups will be conducted with:

Patients with MDD: These discussions will explore their lived experiences with MDD, their perceptions of the overall management of their condition during hospitalization, and their specific experiences with the physical therapy intervention program, including any perceived barriers and facilitators to participation and benefit.

Healthcare Professionals: Focus groups with the multidisciplinary team (including medical, nursing, and other allied health staff) from the short-stay psychiatry unit will focus on their perspectives regarding the integration of physical therapy into the standard care pathway for patients with MDD, their observations of patient engagement and response to the intervention, and any perceived barriers and facilitators to its implementation within the clinical setting.

Focus groups will be guided by semi-structured question guides, audio-recorded with informed consent, and transcribed verbatim. Data collection will continue until thematic saturation is achieved. Thematic content analysis will be employed to identify key patterns and insights from the narratives.

Data Analysis Approach:

The quantitative data, collected at baseline and post-intervention, will be analyzed using appropriate statistical methods for pre-post comparisons in a single group design. Descriptive statistics will summarize the sample characteristics and outcome measures at each time point. Inferential statistics will be used to assess the magnitude and statistical significance of changes in the primary and secondary outcome measures following the intervention.

The qualitative data from the focus groups will be analyzed using thematic content analysis. Transcripts will be independently coded by two researchers, with codes grouped into subcategories and subsequently into overarching themes through a process of iterative refinement and consensus. Measures to ensure the trustworthiness of the qualitative data, such as data and investigator triangulation, will be employed.

Finally, a mixed-methods approach will be used to integrate the quantitative findings on the program's potential efficacy with the rich contextual data obtained from the qualitative component, providing a more comprehensive understanding of the intervention's impact and feasibility.

ELIGIBILITY:
Inclusion and Exclusion Criteria for Patients with Major Depressive Disorder (MDD):

Inclusion Criteria:

* Be 18 years of age or older.
* Be currently admitted to the short-stay inpatient unit of the Psychiatry Department at Royo Villanova Hospital (Zaragoza).
* Have a physician-confirmed diagnosis of Major Depressive Disorder (MDD) according to current diagnostic criteria (ICD-10 or DSM-5).
* Be receiving regular medical, psychological, and/or pharmacological treatment for their MDD.
* Not require continuous supervision and control by nursing staff during data collection and the intervention.
* Have provided written informed consent to participate in the study.

Exclusion Criteria:

* Presence of a comorbid physical or mental illness whose clinical characteristics and/or severity impede comprehension and/or adherence to the physical therapy interventions.
* Presence of a physical or mental dysfunction or disability that constitutes a total or partial contraindication for physical therapy techniques.
* Legal incapacity or pregnancy.
* Present a significant risk of self-harm or suicide requiring clinical management that takes precedence over study participation (this exclusion will be determined by the responsible medical team).

Inclusion and Exclusion Criteria for Healthcare Professionals at Royo Villanova Hospital:

Inclusion Criteria:

* Be a healthcare professional (physician, nurse, physical therapist, occupational therapist, etc.) or non-healthcare staff member (nursing assistant, orderly, etc.) within the short-stay inpatient Psychiatry Department at Royo Villanova Hospital (Zaragoza).
* Be actively employed under a single, permanent, or temporary employment contract throughout the duration of the physical therapy intervention implementation period.
* Have provided written informed consent to participate in the study.

Exclusion Criteria:

* Professionals from the unit who were not actively employed under a single, permanent, or temporary employment contract throughout the entire duration of the physical therapy intervention implementation period.
* Be on sick leave or parental leave during the period of qualitative data collection.
* Have been transferred to another unit or healthcare center prior to the commencement of qualitative data collection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Change in Quality of Life | From enrollment to the end of treatment at 3-6 weeks
  Change in the score on the European quality of life questionnaire or EuroQol 5-Dimension 3-Level Spanish version questionnaire (EQ-5D-3L). The EQ-5D-3L health questionnaire is a questionnaire that can be self-administered or conducted through an interview, which allows for assessing the health status in relation to various patient dimensions (mobility, pain, mental health, etc.). It consists of 5 questions with 3 response options (good health = 1, some problems = 2, or health problem = 3), where the responses are coded and coefficients are applied according to the responses to obtain a reference value; and on the other hand, it consists of a 20-centimeter vertical visual analogue scale, with values from 0 = worst health state to 100 = best health state, where the patient indicates the current perceived health value. It is a validated tool widely used in health and research.

SECONDARY OUTCOMES:
Change in Severity of Depressive Symptoms | From enrollment to the end of treatment at 3-6 weeks
  Change in the score on the Montgomery-Asberg Depression Rating Scale (MADRS) Spanish version. It is a scale used clinically for the detection and severity assessment of major depressive disorder. It consists of 10 questions administered to the interviewee regarding cognitive and affective/emotional symptoms, with response values ranging from 0 to 6 (0 = lowest level of symptomatology and 6 = highest level of symptomatology). Its interpretation is as follows: 0-6 points, no depression; 7-19 points, mild depression; 20-34 points, moderate depression; and 35-60 points, severe depression.
Change in Pain Intensity | From enrollment to the end of treatment at 3-6 weeks
  Change in the score on the Numerical Rating Scale (NRS). The NRS scale for pain assessment is a scale that measures the intensity of pain experienced by the patient. It is a numerical rating scale where the patient is asked to rate their pain between 0 and 10. The reported values are classified as follows: no pain = 0; mild pain = 1,2; moderate pain = 3-5; severe pain = 6-8; unbearable pain = 9-10.
Change in General Self-Efficacy | From enrollment to the end of treatment at 3-6 weeks
  Change in the score on the General Self-Efficacy Scale (GSE) Spanish version. The Spanish version of the General Self-efficacy Scale consists of a 10-item questionnaire that measures an individual's perception of their own abilities to manage their life in stressful situations. For each question, the respondent answers using a Likert scale where the response is scored as 1 = completely disagree and 5 = completely agree. A score between 27 and 38 points is considered an average level of self-efficacy. Higher scores indicate a greater perceived self-efficacy.
Healthcare Satisfaction Level | Up to 6 weeks post-baseline - measured only at this time point
  Score on the Health Care Satisfaction Survey for People with Chronic Illness (GCPC-UN-ESU). It contains 19 items with 4 dimensions: care, health education, the quality of the service provided, and the level of loyalty to the service. Each item is scored between 1 (not at all satisfied) and 5 (extremely satisfied). Higher scores indicate greater satisfaction.

OTHER OUTCOMES:
Focus Group Data: Qualitative Exploration of Patient Experiences and Perceptions in a Physical Therapy Program for Major Depressive Disorder | Following completion of intervention and quantitative assessment up to 6 weeks
  This qualitative outcome measure will use focus groups to explore the experiences and perceptions of patients with major depressive disorder participating in a physical therapy program. Patient narratives will detail their experience with the illness, their condition management strategies, and the barriers and facilitators encountered during the program. Data, collected via audio recordings and field notes from trained researchers, will undergo thematic analysis. Anticipated themes include experiences with physical therapy, perceived impact on symptoms, coping strategies, support systems, adherence factors, facilitators to recovery, and suggestions for program improvement. Qualitative findings will provide context to quantitative results.
Focus Group Data: Qualitative Exploration of Professional Perspectives on Implementing a Physical Therapy Program for Major Depressive Disorder | Within 2 weeks of completion of the quantitative phase
  This qualitative outcome measure will use focus groups to explore the experiences and perspectives of healthcare professionals involved in a physical therapy program for patients with major depressive disorder. Professional narratives will detail their perspectives on managing patients with the illness, their observations of patient condition management strategies, and the barriers and facilitators they encountered during the program's implementation. Data, collected via audio recordings and field notes from trained researchers, will undergo thematic analysis. Anticipated themes include experiences with implementing the physical therapy program, perceived impact on patients, interprofessional collaboration, resource utilization, adherence factors from the professionals' point of view, facilitators to program delivery, and suggestions for program improvement. Qualitative findings will provide context to quantitative results.

CONTACTS AND LOCATIONS:
Overall Officials: Carolina Jiménez Sánchez, Dr, Study Director — Universidad San Jorge; José Lesmes Poveda López, Principal Investigator — Universidad San Jorge
Locations (1):
- Hospital Royo Villanova, Zaragoza, Aragon, Spain

IPD SHARING:
Plan to Share IPD: Yes
All collected individual participant data, including anonymized raw data from questionnaires and clinical assessments, that underlie the results published in any resulting manuscript will be made available.
Supporting Information: Study Protocol
Time Frame: December 2025-July 2026
Access Criteria: Anonymized individual participant data that underlie the results in published manuscripts, including the study protocol and statistical analysis plan, will be made available to researchers who provide a methodologically sound proposal. Proposals should be directed to the corresponding author of the publication. Access will be granted subject to approval by the research team and a data sharing agreement.

REFERENCES:
- [Derived] Poveda-Lopez JL, Jimenez-Sanchez C, Lafuente-Ureta R, Marco-Gomez B, Villagrasa-Cantin A, Perez-Mansilla S, Guarch-Rubio M, Roy JF. Study protocol for a mixed-methods pilot of a physiotherapy plus education program for inpatients with major depressive disorder: Feasibility and preliminary effects. PLoS One. 2025 Nov 6;20(11):e0326012. doi: 10.1371/journal.pone.0326012. eCollection 2025. PMID 41196855